CLINICAL TRIAL: NCT01193894
Title: A Randomized Trial on Profermin and Fresubin for Dietetic Treatment of Active Ulcerative Colitis
Brief Title: Trial on Profermin and Fresubin in Ulcerative Colitis
Acronym: CUPE2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nordisk Rebalance A/S (Industry)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CUPE2
Record Dates: First submitted 2010-08-23; First posted 2010-09-02 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Ulcerative Colitis
Keywords: IBD; UC; Profermin; Fresubin; Probiotics; Dietetic
MeSH Terms: conditions — Colitis, Ulcerative | interventions — profermin; Fresubin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Profermin (Experimental)
  Interventions: Other: Profermin
- Fresubin (Active Comparator)
  Interventions: Other: Fresubin

INTERVENTIONS:
Other: Profermin — Medical Food (food for special medical purposes)
  Arms: Profermin
Other: Fresubin — Medical food (food for special medical purposes)
  Arms: Fresubin

SUMMARY:
This study aim to investigate the effect of Profermin versus Fresubin in the dietetic treatment of active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative colitis (SCCAI =>5 and <=11)
* Access to Internet

Exclusion Criteria:

* Stoma or intestinal resections
* Recent changes in UC medication
* Treatment with antibiotics
* Diabetes
* Celiac disease
* Lactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Development in Simple Clinical Colitis Activity Index (SCCAI) score | 8 and 16 weeks
  Clinical significant difference (>1.5) in course of SCCAI score between the two intervention groups

SECONDARY OUTCOMES:
Reduction in SCCAI score | 8 and 16 weeks
  Proportion of patients with a reduction in SCCAI above 1.5, 3.0 and 4.5
Clinical remission | 8 and 16 weeks
  Proportion of patients in clinical remission (SCCAI=<2.5)
Safety - Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans Israelsen, PhD, Study Director — Nordisk Rebalance A/S; Aleksander Krag, MD, PhD, Principal Investigator — Hvidovre University Hospital; Flemming Bendtsen, MD, DMSci, Study Chair — Hvidovre University Hospital
Locations (1):
- Noreba, Allerød Municipality, Capital Region, Denmark